CLINICAL TRIAL: NCT01642511
Title: Phase II Trail of Internal Mammary Sentinel Lymph Node Biopsy in Early Breast Cancer Patients With Clinically Axillary Node -Negative
Brief Title: Internal Mammary Sentinel Lymph Node Biopsy in Early Breast Cancer Patients With Clinically Axillary Node -Negative
Acronym: IMSLNB-EBCP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Director, Head of Breast Cancer Center, Principal Investigator, Clinical Professor, Shandong Cancer Hospital and Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IMSN001
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Sentinel Lymph Node Biopsy; Internal Mammary; Lymphoscintigraphy
MeSH Terms: conditions — Breast Neoplasms | interventions — Lymphoscintigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): conventional technique: 99mTc-labeled Sulfur Colloid was injected into the tumor quadrant 3-24 hours before surgery, lymphoscintigraphy was performed 30min before surgery. Four milliliters of methylthioninium was injected subcutaneously above the primary tumor or around the biopsy cavity 10 min before surgery. Axillary sentinel lymph node biopsy and Internal mammary sentinel lymph node biopsy was performed during surgery. Axillary lymph node dissection was performed if ASLN was positive.
  Interventions: Radiation: 99mTc-labeled Sulfur Colloid; Procedure: Axillary Sentinel Lymph Node Biopsy; Drug: Methylthioninium; Device: Lymphoscintigraphy; Procedure: Axillary Lymph Node Dissection; Procedure: Internal Mammary Sentinel Lymph Node Biopsy
- Study Group (Experimental): modified technique: 99mTc-labeled Sulfur Colloid was injected into 2 quadrants of the breast 3-24 hours before surgery, lymphoscintigraphy was performed 30min before surgery. Four milliliters of methylthioninium was injected subcutaneously above the primary tumor or around the biopsy cavity 10 min before surgery. Axillary sentinel lymph node biopsy and Internal mammary sentinel lymph node biopsy was performed during surgery. Axillary lymph node dissection was performed if ASLN was positive.
  Interventions: Procedure: Axillary Sentinel Lymph Node Biopsy; Drug: Methylthioninium; Device: Lymphoscintigraphy; Procedure: Axillary Lymph Node Dissection; Procedure: Internal Mammary Sentinel Lymph Node Biopsy

INTERVENTIONS:
Radiation: 99mTc-labeled Sulfur Colloid — Control Group: Each patient received the 1 intraparenchymal injection of 99mTc-SC (0.5~1.0 mCi/0.5mL) in the tumor quadrant. Study Group: Two syringes of 0.25~0.5 mCi 99mTc-SC in 0.2~1.0 mL volume were injected intraparenchymally into 2 quadrants of breast, at the 6 and 12 o'clock positions.
  Other Names: 99mTc-SC
  Arms: Control Group
Procedure: Axillary Sentinel Lymph Node Biopsy — Sentinel lymph node biopsy
  Other Names: SLNB
Drug: Methylthioninium — Four milliliters of methylthioninium was injected subcutaneously above the primary tumor or around the biopsy cavity 10 min before surgery
Device: Lymphoscintigraphy — Sequential anterior and lateral gamma imaging was performed with patients lying prone and by injection side just before surgery using a digital gamma camera computer system (Toshiba GCA-901A/HG).
  Other Names: LSG
Procedure: Axillary Lymph Node Dissection — ALND was performed consequently if axillary SLNB was failure or axillary SLNs were positive.
  Other Names: ALND
Procedure: Internal Mammary Sentinel Lymph Node Biopsy — Internal mammary sentinel lymph node biopsy
  Other Names: IM-SLNB

SUMMARY:
In addition to the axillary lymph node, the internal mammary lymph node (IMLN) chain is also the first-echelon nodal drainage site for metastasis and provides important prognostic information in breast cancer patients. The internal mammary sentinel lymph node biopsy (IM-SLNB) provides a less invasive method of assessing the IMLN than surgical dissection. But the low visualization rate of IMSLN has been a restriction of IM-SLNB. This clinical trial is carried out to improve the visualization rate of IMSLN with modified techniques: (1) The radiotracer is injected intraparenchymally into 2~4 quadrants of breast. (2) The radiotracer is injected in a high volume. (3) The radiotracer should be injected under ultrasonographic guidance.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the visualization rate of internal mammary sentinel lymph node in breast cancer patients with different injection technologies.
* Evaluate the metastasis rate of internal mammary sentinel lymph nodes in patients with clinically axillary node -negative in these patients.
* Evaluate the risk factors for internal mammary sentinel lymph node metastasis
* Evaluate the success rate and the safety of internal mammary sentinel lymph node biopsy.
* Draw the learning curve of internal mammary sentinel lymph node biopsy.

OUTLINE:

3~18 hours before surgery, 99mTc-labeled sulfur colloid was injected under ultrasonographic guidance in different patterns and injection methods were classified according to the number of injection quadrants. Subsequently, lymphoscintigraphy was performed 0.5~1.0 hour before surgery. During surgery, the sentinel lymph nodes (axillary or internal mammary) were identified by combining the use of intraoperative gamma detector and blue dye. The sentinel lymph nodes (axillary or internal mammary) were analyzed by hematoxylin-eosin staining and immunohistochemistry for future therapy planning.

ELIGIBILITY:
Inclusion Criteria:

* primary breast cancer
* clinically axilla-negative

Exclusion Criteria:

* enlarged internal mammary nodes by imaging

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Visualization rate of IMSLN | 1 year
  Visualization rate of IMSLN between conventional and modified techniques

SECONDARY OUTCOMES:
Metastasis Rate of IMSLN | 15 months
  Metastasis rate of IMSLN in clinically axillary node-negative patients with IM-SLNB
Frequency and Severity of Complications with IM-SLNB | 1 year
  IM-SLNB complications in the patients who receive IM-SLNB
Success rate of IM-SLNB | 1 year
  Success rate of IM-SLNB in the IMSLN visualization patients who receive IM-SLNB

CONTACTS AND LOCATIONS:
Overall Officials: Yong-sheng Wang, MD, Study Chair — Shandong Cancer Hospital and Institute; Peng-fei Qiu, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China

REFERENCES:
- [Result] Qiu PF, Liu JJ, Liu YB, Yang GR, Sun X, Wang YS. A modified technology could significantly improve the visualization rate of the internal mammary sentinel lymph nodes in breast cancer patients. Breast Cancer Res Treat. 2012 Nov;136(1):319-21. doi: 10.1007/s10549-012-2203-5. Epub 2012 Sep 6. No abstract available. PMID 22956005
- [Derived] Qiu P, Zhao R, Cong B, Yang G, Liu Y, Chen P, Sun X, Wang C, Wang Y. [Internal mammary sentinel lymph node biopsy in breast cancer: accurate staging and individualized treatment]. Zhonghua Zhong Liu Za Zhi. 2016 Jan;38(1):42-7. doi: 10.3760/cma.j.issn.0253-3766.2016.01.009. Chinese. PMID 26796806